CLINICAL TRIAL: NCT05829057
Title: The IIT Study of Evaluation of Platelet-coupled IL-2 Cell Injection (P-IL-2) Single Agent and With Anti-PD-1 Monoclonal Antibody on the Safety, Tolerance and Preliminary Effectiveness in Patients With Advanced Malignant Solid Tumors
Brief Title: The IIT Study of Evaluation of P-IL-2 Single Agent and With Anti-PD-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Zcapsule Pharmaceuticals (Shaoxing) Co., Ltd (Industry)
Responsible Party: Principal Investigator, Weijia Fang, MD, Principal Investigator, Zhejiang University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZS205
Record Dates: First submitted 2023-03-14; First posted 2023-04-25 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Esophagus Cancer; Bladder Cancer; Liver Cancer; Ovarian Cancer; Small-cell Lung Cancer
Keywords: cancer
MeSH Terms: conditions — Esophageal Neoplasms; Urinary Bladder Neoplasms; Liver Neoplasms; Ovarian Neoplasms; Small Cell Lung Carcinoma; Neoplasms

STUDY DESIGN:
Intervention Model Description: Arms and Interventions： Experimental: Arm of P-IL-2 Based on platelet count： Cohort 1：8×10^9 PLT； Cohort 2：2.5×10^10 PLT； Cohort 3：8×10^10 PLT； Cohort 4：2.5×10^11 PLT/kg BW； Experimental: P-IL-2 plus Anti-PD-1 Monoclonal Antibody
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm of P-IL-2 (Experimental): Ia:Subjects will be dosed with single dose of P-IL-2
  Interventions: Biological: Intravenous injection of P-IL-2
- P-IL-2 plus Anti-PD-1 Monoclonal Antibody (Experimental): Ib:Subjects will be dosed with dose of P-IL-2 plus Anti-PD-1 Monoclonal Antibody
  Interventions: Biological: P-IL-2 plus Anti-PD-1 Monoclonal Antibody

INTERVENTIONS:
Biological: Intravenous injection of P-IL-2 — Ia :Single dose intravenous injection of P-IL-2；
  Arms: Arm of P-IL-2
Biological: P-IL-2 plus Anti-PD-1 Monoclonal Antibody — Ib：P-IL-2 plus Anti-PD-1 Monoclonal Antibody；
  Arms: P-IL-2 plus Anti-PD-1 Monoclonal Antibody

SUMMARY:
Phase Ia: single-dose escalation study: accelerated titration combined with traditional "3+3" dose. Sample size is correlated with the DLT occurring in each dose group. 4 dose groups are expected; the first dose group is the accelerated titration group, which includes only 1 subject; subsequent dose groups are in traditional "3+3" dose increments, with 3-6 subjects in each group; a total of 10-19 subjects are expected in all dose groups. If the DLT is still not present in the highest dose ,the safety monitoring committee(SMC) to determine if it is necessary to continue incrementally to a higher dose.

DETAILED DESCRIPTION:
P-IL-2 injection was injected intravenously, the screening period was 28 days, and the DLT observation period was 28 days from the beginning of the first infusion (including the day of administration). After the end of the DLT observation period, subjects can continue to receive treatment on a voluntary basis. The safety follow-up after drug withdrawal was carried out 28 days after the last medication. During the survival follow-up after drug withdrawal, imaging examination and survival information were collected every 12 weeks as far as possible within 2 years after drug withdrawal, until the subjects developed disease or received other anti-tumor specific therapy. Subjects with disease progression or other treatment received telephone survival follow-up every 12 weeks. After 2 years of drug withdrawal, telephone survival follow-up was conducted every 12 weeks according to the wishes of the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to follow study procedures , and sign a written informed consent form;
2. Males or females aged 18-75 years old at the time of signing the ICF;
3. Expected survival time ≥ 12 weeks.
4. Physical condition score ECOG ≤ 1.
5. There is still disease progression, intolerance or lack of effective standard treatment under standard treatment. Patients with advanced malignant solid tumor confirmed by pathology (recurrence and / or metastasis); at least 1 Measurable lesions in accordance with RECIST v1.1 or iRECIST standards.
6. Before the first administration, it had recovered from the toxic effects of the last treatment, and the researchers determined that the corresponding AE did not have a safety risk.
7. Organ and bone marrow function levels must meet the following requirements:

   Bone marrow: absolute neutrophil count (ANC) ≥ 1.5 × 109 ppm L, specified value (according to Group determination, see Appendix 11 for instructions on platelet count during the screening period), platelets Count ≥ 100x109 shock L, hemoglobin ≥ 90g/L, and no blood transfusion within 14 days before the first administration.
8. Male subjects and female subjects of childbearing age from the signing of informed consent form to the end of drug research. Voluntary use of effective contraceptive measures within 5 months after secondary use.

Exclusion Criteria:

1. Past or present suffering from other types of malignant tumors.
2. Known to be allergic to research drugs or any of their excipients, or to be too strict with other monoclonal antibodies.Severe anaphylaxis (NCI-CTCAE 5.0 grade ≥ 3).
3. People have hemorrhagic diseases or have hemorrhagic tendencies.
4. Received any of the following treatments or drugs before the first study:

   * large surgery or severe trauma occurred within 4 weeks before the first study of drug treatment.
   * previous use of immunosuppressive drugs within 2 months prior to the first study, excluding nasal spray.
   * And inhaled corticosteroids or physiological doses of systemic steroids.
   * to study the Chinese medicine therapy with anti-tumor indications within 2 weeks before drug treatment for the first time.
5. Patients with a history of central nervous system metastasis (non-tumor meningeal metastasis) or spinal cord compression can be enrolled in the study if they have clearly received treatment and have stopped taking anticonvulsants and steroids for 4 weeks or more and have stable clinical manifestations before the first administration of the study.
6. Symptomatic, visceral spread, and short-term risk of life-threatening complications. the patients who underwent puncture and drainage within 3 weeks before the first administration included pleural effusion and abdominal cavity. Patients with effusion and pericardial effusion.
7. Subjects with active, or history of autoimmune diseases that may recur, or patients at high risk. subjects with the following diseases are allowed to join the group:

   * stable type I diabetic patients treated with fixed dose of insulin.
   * autoimmune hypothyroidism which only needs hormone replacement therapy.
   * skin diseases that do not require systemic treatment.
   * cured childhood asthma / allergy adult patients without any intervention.
8. Within 6 months before screening, any cardiovascular disease met any of the following criteria:

   * congestive heart failure with heart function ≥ New York Heart Association (NYHA) Class II; left ventricular ejection. Blood fraction (LVEF) < 50%.
   * severe arrhythmias requiring drug treatment.
   * QTcF (Fridericia formula) male > 450ms, female > 470ms, or exist risk factors of apical torsion ventricular tachycardia are of clinical significance .
   * myocardial infarction and severe / unstable angina pectoris occurred within 6 months before administration.
   * history of thromboembolism with grade 3 or more in the past 2 years, or is being received because of a high risk of thrombosis.

   Receive thrombolytic or anticoagulant therapy.
9. Currently suffering from sudden lung disease, interstitial lung disease or pneumonia, pulmonary fibrosis, acute lung disease, etc., except local interstitial pneumonia caused by radiotherapy.
10. Uncontrolled systemic diseases .
11. history of human immunodeficiency virus infection, or suffer from other acquired, congenital immunodeficiency. Disease, or a history of organ transplantation, or a history of stem cell transplantation;
12. Evidence of active infection.
13. Previous history of neurological or mental disorders, or known history of psychotropic substance abuse and alcoholism.

    History or history of drug use.
14. Received any research drug within 4 weeks before the first administration, or participated in another clinical trial at the same time.
15. Female patients who are pregnant or lactating, or whose baseline pregnancy test results are positive.
16. The researchers believe that it is not suitable for patients to be included in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-21 (Estimated)

PRIMARY OUTCOMES:
the number and severity of DLTs. | 28 days after infusion
  DLT refers to toxicities that occur within 28 days of the subject's first dose and are judged by the investigator to be related to the study drug and meet the following conditions, including any ≥4 hematologic toxicity and non-hematologic toxicity. All toxicity or adverse events (AEs) are graded according to NCI-CTCAE 5.0.
Incidence of AE and SAE | 24 month after infusion
  Incidence and Severity of AE and SAE; An AE was any untoward medical occurrence after clinical study subjects receive study drug. An SAE was any event that meets any the following criteria: death, life-threatening; inpatient hospitalization or prolongation, persistent or significant disability/incapacity; congenital malformation/birth defects and significant medical events. AE and SAE were graded by CTCAE version 5.0 by severity, from Grade 1 mild to Grade 5 death related AE.
Number of participants with physical examinations | 24 months after infusion
  Make list of patients who were normal before administration and abnormal after administration, physical examinations includes general appearance and examinations of the skin, eyes, ears, nose, throat, lungs, heart, abdomen, limbs, musculoskeletal system, nervous system and lymphatic system.

SECONDARY OUTCOMES:
changes in the number of CD3+ cells relative to the baseline. | Within 28 days after infusion
  Peripheral blood collection, number of CD3+ cells is detected by qPCR
changes of immunoglobulin IgG relative to the baseline. | Within 28 days after infusion
  Peripheral blood collection, to monitor the changes of IgG
changes of immunoglobulin IgE relative to the baseline. | Within 28 days after infusion
  Peripheral blood collection, to monitor the changes of IgE
changes of cytokines relative to the baseline | Within 28 days after infusion
  Peripheral Blood collection，cytokines include IFN-γ、TNF-α、IL-2、IL-6、IL-10

CONTACTS AND LOCATIONS:
Overall Officials: weijia weijia, Principal Investigator — stem cell and somatic cell clinical study committee
Locations (1):
- First affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No